CLINICAL TRIAL: NCT02937935
Title: On Demand Versus Protocol-guided Renal Replacement Therapy for Management of Stage 3 Acute Kidney Injury in Patients With Cirrhosis -A Prospective Randomized Controlled Trial
Brief Title: On Demand Versus Protocol-guided Renal Replacement Therapy for Management of Stage 3 Acute Kidney Injury in Patients With Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AKI-Cirrhosis
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Acute Kidney Injury With Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol Guided-RRT (Experimental): In the on-demand group patients would get dialysis only when patient fulfills absolute criteria requiring dialysis such as metabolic acidosis with ph<7.2, hyperkalemia, refractory fluid overload (non-responsive to diuretics) or oliguria with urine output of less than 0.5ml/kg for more than 24-48 hours from the time of randomization.
  Interventions: Biological: Protocol Guided Renal Replacement Therapy
- On Demand-RRT (Active Comparator): In the protocol guided group patients all patients would be considered for dialysis within 6 hours of randomization After randomization patients would receive dialysis as three sessions per week of at least 4 h with a blood flow >200 mL/min and a dialysate flow >500 mL/min in intermittent group and as 20-25 mL/kg/h of effluent, by filtration and/or diffusion in continuous form until recovery of renal functions
  Interventions: Biological: On Demand Renal Replacement Therapy

INTERVENTIONS:
Biological: Protocol Guided Renal Replacement Therapy — In the on-demand group patients would get dialysis only when patient fulfills absolute criteria requiring dialysis such as metabolic acidosis with ph<7.2, hyperkalemia, refractory fluid overload (non-responsive to diuretics) or oliguria with urine output of less than 0.5ml/kg for more than 24-48 hours from the time of randomization.
  Arms: Protocol Guided-RRT
Biological: On Demand Renal Replacement Therapy — Patients to be randomized to the intervention as per standard of care
  Arms: On Demand-RRT

SUMMARY:
Intervention: All patients at presentation would be assessed for the underlying cause of and will be managed by removal of all precipitants(careful review of medications, diuretics, nephrotoxic drugs,vasodilators or non-steroidal anti-inflammatory drugs). The second step would be to consider plasma volume expansion in patients with hypovolemia (the choice of fluid could either be a crystalloid or albumin or even blood as indicated) along with identification and early treatment of bacterial infections. Along with this patients with a differential diagnosis of HRS-AKI would be given terlipressin ( or noradrenaline/octreotide midodrine in case of contraindication to terlipressin). Patients with a clinical diagnosis of ATN would be randomized to the on-demand versus protocol-guided dialysis groups. Further, patients with urine output of less than 0.5ml/kg/hour for 4-6 hours despite adequate fluid resuscitation and vasoconstrictors would also be subjected to randomization.

1. In the on-demand group patients would get dialysis only when patient fulfills absolute criteria requiring dialysis such as metabolic acidosis with ph<7.2, hyperkalemia, refractory fluid overload (non-responsive to diuretics) or oliguria with urine output of less than 0.5ml/kg for more than 24-48 hours from the time of randomization
2. In the protocol guided group patients all patients would be considered for dialysis within 6 hours of randomization After randomization patients would receive dialysis as three sessions per week of at least 4 h with a blood flow >200 mL/min and a dialysate flow >500 mL/min in intermittent group and as 20-25 mL/kg/h of effluent, by filtration and/or diffusion in continuous form until recovery of renal functions

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis (diagnosed based on clinical, biochemical,radiological or histological diagnosis) with stage 3 Acute Kidney Injury defined as an increase of serum creatinine to more than 300 fold and more than 4 mg/dl.

Exclusion Criteria:

* Patients with age less than 18 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD Chronic Obstructive Pulmonary Disease)
* Pregnancy
* Chronic kidney disease on hemodialysis
* Patients with post renal obstructive AKI (Acute Kidney Injury), AKI (Acute Kidney Injury) suspected due to glomerulonephritis, interstitial nephritis or vasculitis based on clinical history and urine analysis
* Patients already meeting emergency criteria for immediate hemodialysis at the time of randomization (serum potassium>6 meq/lt, metabolic acidosis ph<7.12, acute pulmonary edema, severe volume overload with hypoxemia non-responsive to diuretic treatment)
* Patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Hemodynamic instability requiring very high dose of vasopressors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Recovery of renal functions in both groups | day 14

SECONDARY OUTCOMES:
Adverse effects of dialysis in the first session in both groups | 48 hours
Improvement in SOFA (by 2 points) scores in both groups | 48 hours
Improvement in MELD ( by 2 points) scores in both groups | 48 hours
Improvement in APACHE ( by 2 points) scores in both groups | 48 hours
Change to End Stage Renal Disease with requirement of maintenance hemodialysis at least twice a week in both groups | 4 weeks
Improvement in renal functions in both groups | 7 days
Mortality in both groups | 1 month
Mortality in both groups | 3 month
Response to vasoconstrictors in patients with Hepatorenal Syndrome-Acute Kidney Injury in both groups. | 6 hours
  Response as assessed by either improvement in urine output >0.5ml/kg/hour, acid-base status or renal functions.
Response to vasoconstrictors in patients with Hepatorenal Syndrome-Acute Kidney Injury in both groups. | 12 hours
  Response as assessed by either improvement in urine output >0.5ml/kg/hour, acid-base status or renal functions.
Response to vasoconstrictors in patients with Hepatorenal Syndrome-Acute Kidney Injury | 24 hours
  Response as assessed by either improvement in urine output >0.5ml/kg/hour, acid-base status or renal functions.
Response to vasoconstrictors in patients with Hepatorenal Syndrome-Acute Kidney Injury in both groups | 24 hours
  Response as assessed by either improvement in urine output >0.5ml/kg/hour, acid-base status or renal functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787